CLINICAL TRIAL: NCT02477319
Title: A Two-Part Multicenter Prospective Longitudinal Study of CFTR-dependent Disease Profiling in Cystic Fibrosis (PROSPECT)
Acronym: PROSPECT
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: PROSPECT
Record Dates: First submitted 2015-05-22; First posted 2015-06-22 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part A: * Cohort 1: Healthy Controls
  * Cohort 2: Partial CFTR function CF (class IV/V)
  * Cohort 3: Absent CFTR function CF (Class I/II)
  Interventions: Other: Observational
- Part B: CF patients who are homozygous for the F508del
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
identify and validate biomarkers that might reflect partial restoration of CFTR function and can be used to monitor disease progression, and ii) evaluate the mechanistic effects of CFTR modulators and other relevant therapies in individuals with CF

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disorder caused by mutations in the gene encoding the cystic fibrosis transmembrane conductance regulator (CFTR) protein. Over 1,900 mutations, categorized into five genotypic or functional classes are implicated in causing CF. Severity of disease varies widely in CF based on CFTR-dependent and independent factors. Progressive obstructive lung disease is the main determinant of morbidity and mortality in CF; therefore it is critical to identify biomarker profiles that reflect and predict this phenotypic variability, and understand their relationship to residual CFTR activity. Emerging CFTR modulator therapies that directly target defective CFTR are being evaluated in pivotal clinical trials and may become available in the next few years. It is not known how partial restoration of CFTR function might impact CF disease progression and disease-related biomarkers. Thus there is urgent need to i) identify and validate biomarkers that might reflect partial restoration of CFTR function and can be used to monitor disease progression, and ii) evaluate the mechanistic effects of CFTR modulators and other relevant therapies in individuals with CF

ELIGIBILITY:
Inclusion Criteria Part A COHORT 1:

* 1. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.

  2. Be willing and able to adhere to the study visit schedule and other protocol requirements 3. Male or female ≥ 12 years of age at Visit 1. 4. Have a body mass index (BMI) of:
  * For subjects ≥ 18 years of age: ≤ 30 kg/m2
  * For subjects 12 - 17 years of age: ≤ 95th percentile 5. Be a non-smoker for ≥ 1 year at screening and have ≤ 10 pack-year history of smoking.

    6. To participate in the optional DNA banking component of this study, subject must have signed the informed consent indicating willingness to participate in the genomic component of the study. Refusal to give consent for this component does not exclude a subject from participation in the study.

Inclusion Cohorts 2-3

1. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.
2. Male or female ≥ 12 years of age at Visit 1.
3. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and the following criteria: Cohort 2: (Partial Function CFTR CF)

   * Two mutations in the CFTR gene:

     * At least one allele must be a Class IV or V mutation
     * The second allele can be within any CFTR mutation class.
   * Pancreatic sufficient (based on the absence of daily PERT use)
   * At least one historic sweat chloride ≥60 mEq/L by quantitative pilocarpine iontophoresis test (QPIT) OR sweat chloride results ≥ 40, but < 60mEQ/L upon permission of the PROSPECT Investigator-Sponsors.

   Cohort 3: (Absent Function CF)

   • Two class I or II CFTR mutations
4. Enrolled in the Cystic Fibrosis Foundation Patient Registry. Patients may enroll in the Registry at Visit 1 if not previously enrolled.
5. Clinically stable with no significant changes in health status within 2 weeks prior to Visit 1.
6. Be a non-smoker for ≥ 1 year at screening and have ≤ 10 pack-year history of smoking.
7. To participate in the optional DNA banking component of this study, subject must have signed the informed consent indicating willingness to participate in the genomic component of the study. Refusal to give consent for this component does not exclude a subject from participation in the study

Part B Inclusion

1. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative.
2. Physician decision to treat with ivacaftor/lumacaftor.
3. Completion of at least Visit 1 and Visit 2 of Part A

Exclusion Criteria PART A COHORT 1

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. A history of any clinically significant medical illness or medical disorder that requires ongoing systemic medical therapy, including (but not limited to) cardiovascular disease, neuromuscular disease, hematological disease including bleeding disorders, chronic respiratory disease (including persistent asthma), hepatic or gastrointestinal (GI) disease, neurological disease, neoplastic disease, renal diseases, or endocrine disorders including diabetes.
3. Acute illness requiring any new prescription or over-the-counter treatment within 14 days prior to Visit 1.
4. Major or traumatic surgery within 12 weeks prior to Visit 1.
5. For females of child-bearing potential: a positive pregnancy test at Visit 1.
6. Initiation of any new chronic therapy within 28 days prior to Visit 1.
7. Use of an investigational agent within 28 days prior to Visit 1.

Exclusion Part A COHORTS 2-3

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Initiation of newly prescribed antibiotics [oral, intravenous (IV), and/or inhaled] for acute respiratory symptoms within 2 weeks of Visit 1.
3. Major or traumatic surgery within 12 weeks prior to Visit 1.
4. For females of child-bearing potential: a positive pregnancy test at Visit 1.
5. Initiation of any new chronic therapy (e.g., ibuprofen Pulmozyme®, hypertonic saline, azithromycin, TOBI®, Cayston®) within 4 weeks prior to Visit 1.
6. Use of an investigational agent within 28 days prior to Visit 1.
7. Use of oral corticosteroids in doses exceeding 10 mg prednisone/day or 20 mg prednisone/every other day (subjects on oral steroids will be on stable doses for > 12 weeks prior to visit 1).
8. Active treatment for nontuberculous mycobacterial (NTM) infection, consisting of ≥ two antibiotics (oral, IV, and/or inhaled).
9. Use of CFTR modulator therapy such as ivacaftor (Kalydeco®) within 28 days prior to Visit 1.
10. History of lung or liver transplantation, or listing for organ transplantation.

Exclusion PART B

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
2. Initiation of newly prescribed antibiotics [oral, intravenous (IV), and/or inhaled] for acute respiratory symptoms within 2 weeks of Visit 4.
3. Initiation of any new chronic therapy (e.g., ibuprofen, Pulmozyme®, hypertonic saline, azithromycin, TOBI®, Cayston®) within 4 weeks prior to Visit 4.
4. Use of an investigational agent within 28 days prior to Visit 4.
5. Use of oral corticosteroids in doses exceeding 10 mg prednisone/day or 20 mg prednisone/every other day (subjects on oral steroids will be on stable doses for > 12 weeks prior to Visit 4).
6. Active treatment for nontuberculous mycobacterial (NTM) infection, consisting of ≥ two antibiotics (oral, IV, and/or inhaled).
7. Use of CFTR modulator therapy such as ivacaftor (Kalydeco®) within 28 days prior to Visit 4.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Part A N = 260 (210 CF, 50 non-CF controls)
  * Cohort 1: 50 non-CF control subjects ≥ 12 years of age, with at least 15 subjects 12 - 21 yrs of age
  * Cohort 2: 50 Partial CFTR Function CF subjects with at least one class IV/V CFTR mutation, ≥ 12 years of age
  * Cohort 3 160 Absent CFTR Function CF subjects with two class I/II mutations ≥ 12 years of age
  Part B
  Up to 250 CF subjects who are homozygous for F508del mutation and who are prescribed ivacaftor/lumacafor for clinical care will be allowed to enroll. This will include :
  * Cohort 3 subjects homozygous for F508del mutation from Part A who are prescribed ivacaftor/lumacaftor will be invited to participate in Part B (up to 100 potential subjects).
  * Up to 150 additional CF subjects homozygous for F508del mutation ≥ 12 years of age who did not participate in Part A but are otherwise eligible for participation in Part B.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04-25 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile S. Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital Colarado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indianapolis University Hospital; James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - The University of Kansas Hospital, Kansas City, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Devon Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Maria Fareri Children's Hospital; Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Nation Wide Childrens Hospital, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center; Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sagel SD, Khan U, Heltshe SL, Clancy JP, Borowitz D, Gelfond D, Donaldson SH, Moran A, Ratjen F, VanDalfsen JM, Rowe SM. Clinical Effectiveness of Lumacaftor/Ivacaftor in Patients with Cystic Fibrosis Homozygous for F508del-CFTR. A Clinical Trial. Ann Am Thorac Soc. 2021 Jan;18(1):75-83. doi: 10.1513/AnnalsATS.202002-144OC. PMID 32644818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: March 2015 - June 2017 (revised)
Groups:
- Part A (Cohort 1): • Cohort 1: Healthy Controls
  Observational
- Part A (Cohort 2): Cohort 2: Partial CFTR function CF (class IV/V)
  Observational
- Part A (Cohort 3): Cohort 3: Absent CFTR function CF (Class I/II)
  Observational
- Part B: F508del homozygous CF patients who initiated Lumacaftor/Ivacaftor
  Observational (pre/post study)
Period: Overall Study
Arm/Group | Part A (Cohort 1) | Part A (Cohort 2) | Part A (Cohort 3) | Part B
Started | 55 | 40 | 164 | 193
Completed | 55 | 37 | 149 | 171
Not Completed | 0 | 3 | 15 | 22

BASELINE CHARACTERISTICS:
Groups:
- Part A (Cohort 2): • Cohort 2: Partial CFTR function (CF class IV/V)
  Observational
- Part A (Cohort 3): • Cohort 3: Absent CFTR function (CF Class I/II)
- Total: Total of all reporting groups
Arm/Group | Part A (Cohort 1) | Part A (Cohort 2) | Part A (Cohort 3) | Part B | Total
Number analyzed (Participants) | 55 | 40 | 164 | 193 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (10.1) | 32.3 (18.1) | 21.8 (9.6) | 19.0 (10.6) | 22.0 (11.7)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: >=6 - 11 Y | 0 | 0 | 0 | 45 | 45
  Age Category: >= 12 - 17 | 13 | 11 | 77 | 72 | 173
  Age Category: >= 18 - 29 | 30 | 13 | 53 | 42 | 138
  Age Category: >= 30 | 12 | 16 | 34 | 34 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 84 | 106 | 240
  Male | 29 | 16 | 80 | 87 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 6 | 0 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 0 | 7
  White | 42 | 38 | 155 | 189 | 424
  More than one race | 3 | 0 | 6 | 2 | 11
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
FEV1 % Predicted [Mean (Standard Deviation); unit: % Predicted] — FEV1 % Predicted based on Global Lung Initiative (GLI) equations Population: Cohort 1 participants did not perform spirometry procedures (i.e. are missing baseline FEV1 % Predicted). Also, one Cohort 2 participant is missing baseline spirometry.
  % Predicted
    number analyzed (Participants) | 0 | 39 | 164 | 193 | 396
    (all) |  | 86.9 (24.6) | 81.8 (23.4) | 85.0 (22.4) | 83.9 (23.1)

OUTCOME MEASURES:

1. Primary Outcome: Sweat Chloride by Cohort (Part A Only)
Description: This is the primary endpoint for Part A per the PROSPECT protocol. Mean sweat chloride was not reported for Part B, as it is not a relevant statistic.
  For cohort 1, sweat chloride is from day 0 only. For cohorts 2-3, sweat chloride was averaged from days 0, 14, 90 via a random intercept longitudinal model.
Time Frame: For cohort 1, sweat chloride at Day 0 is time frame. For cohorts 2-3, sweat chloride averaged across all 3 visits at days 0, 14 and 90 is time frame.
Population: Participants with Sweat Chloride measure. For Cohort 1, sweat chloride was collected at Visit 1 only (Day 0). Cohort 2 and 3 were collected at Days 0, 14 and 90.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Part A (Cohort 1): Cohort 1: Healthy Controls Observational
- Part A (Cohort 2): Cohort 2: Partial CFTR function (CF class IV/V)
- Part A (Cohort 3): Cohort 3: Absent CFTR function (CF class I/II)
Arm/Group | Part A (Cohort 1) | Part A (Cohort 2) | Part A (Cohort 3)
Number analyzed (Participants) | 53 | 40 | 162
mmol/L | 22.0 [19.2 to 24.7] | 81.0 [74.3 to 87.7] | 101.4 [100.1 to 102.7]

2. Primary Outcome: 6 Month Change in FEV1 Percent Predicted (Part B Only)
Description: This is the primary endpoint for Part B per the PROSPECT protocol. Change in FEV1 Percent Predicted is only relevant for Part B as it captures changes in lung function post-initiation of Ivacaftor/Lumacaftor.
Time Frame: Baseline and 6 months
Population: Change in FEV1 % predicted was measured in all participants who had baseline visit and 6 month visit.
Measure: Mean (95% Confidence Interval); unit: Percent Predicted
Groups:
- Part B: Participants who initiated Ivacaftor/Lumacaftor
Arm/Group | Part B
Number analyzed (Participants) | 176
Percent Predicted | -0.2 [-1.7 to 1.2]

ADVERSE EVENTS:
Time Frame: [Not Specified]
Description: This was an observational study. Adverse events were not an endpoint.
Groups:
- All Arms/Groups: Adverse Events were not analyzed by Arm/Group.
Arm/Group | All Arms/Groups
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02477319/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT02477319/SAP_001.pdf